CLINICAL TRIAL: NCT03029403
Title: A Phase 2 Study of Pembrolizumab (MK-3475), DPX-Survivac Vaccine and Low Dose of Cyclophosphamide Combination in Patients With Advanced Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Phase 2 Study of Pembrolizumab, DPX-Survivac Vaccine and Cyclophosphamide in Advanced Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PESCO
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer; Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation (Experimental): Patients with epithelial ovarian, fallopian tube or primary peritoneal cancer.
  Interventions: Drug: Pembrolizumab; Biological: DPX-Survivac; Drug: Cyclophosphamide
- Dose Expansion - Cohort A (Experimental): Patients with platinum-sensitive epithelial ovarian, fallopian tube or primary peritoneal cancer.
  Interventions: Drug: Pembrolizumab; Biological: DPX-Survivac; Drug: Cyclophosphamide
- Dose Expansion - Cohort B (Experimental): Patients with platinum-resistant epithelial ovarian, fallopian tube or primary peritoneal cancer.
  Interventions: Drug: Pembrolizumab; Biological: DPX-Survivac; Drug: Cyclophosphamide
- Dose Expansion - Cohort C (Experimental): Patients with recurrent advanced epithelial ovarian, fallopian tube and primary peritoneal patients with uncommon tumor histologies, including clear cell, mucinous and low grade serous or low grade endometrioid ovarian subtypes.
  Interventions: Drug: Pembrolizumab; Biological: DPX-Survivac; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pembrolizumab — Given intravenously in clinic, at 200 mg, on Day 1 of every 21-day cycle.
  Other Names: Keytruda
Biological: DPX-Survivac — Given by injection under the skin of the upper thigh in clinic. Participants will receive one priming dose of 0.25 mL of DPX-Survivac on Cycle 1 Day 1. After about 6 weeks, participants will receive an additional boosting dose of 0.25 or 0.5 mL DPX-Survivac.
Drug: Cyclophosphamide — Given orally, at 50 mg, twice a day, starting about 7 days before Cycle 1 Day 1, then continue 7 days off, 7 days on.
  Other Names: Procytox

SUMMARY:
This is a phase 2 study whose purpose is to see whether the combination of of pembrolizumab, DPX-Survivac vaccine and low-dose cyclophosphamide has anti-tumor activity in patients with advanced epithelial ovarian, fallopian tube or primary peritoneal cancer.

DPX-Survivac is an investigational vaccine. A vaccine is a substance that is often given to stimulate the body's immune system (the structure and processes in the body that protects against harmful substances) to help prevent against certain diseases. DPX-Survivac is a vaccine that may teach the immune system to recognize cancer cells and to kill them.

Pembrolizumab is a drug that is approved for the treatment of a certain type of melanoma (a type of skin cancer) and non-small cell lung cancer. Pembrolizumab blocks the function of a protein called programmed cell death receptor-1 (PD-1). PD-1 works by keeping the immune system from destroying cancer cells. Stopping PD-1 from working may help the immune system to fight cancer cells.

Cyclophosphamide is chemotherapy drug that is approved for the treatment of various cancers alone and in combination with other drugs.

DETAILED DESCRIPTION:
This study has two phases: a dose escalation phase and a dose expansion phase.

For the dose escalation part, groups of participants will receive one of two dose levels of study drugs to determine the best dose level for further testing.

Once the best dose level is found, additional participant will be enrolled to the dose expansion to further test the safety, tolerability, and efficacy of the study drugs at that dose level in specific types of cancers. All participants will receive pembrolizumab, DPX-Survivac, and low-dose cyclophosphamide.

Participants will be screened for eligibility by standard safety tests and procedures within 28 days of the start of the study drug. Tests and procedures done for research purposes only during this time include archival tumor tissue collection, fresh research biopsy, and blood sample collection for biomarker/genetic/immune research. Participants will also be asked if they agree to an optional fresh research biopsy at disease progression

Eligible participants will receive the following every 21 day cycle:

* Pembrolizumab, intravenously, at 200 mg, on Day 1 of every cycle.
* DPX-Survivac, by injection under the skin of the upper thigh in clinic. Participants will receive one priming dose of 0.25 mL of DPX-Survivac on Cycle 1 Day 1. After about 6 weeks, participants will receive an additional boosting dose of 0.25 or 0.5 mL DPX-Survivac depending on the assigned dose level.
* Cyclophosphamide, orally, at 50 mg, twice a day, starting about 7 days before Cycle 1 Day 1, then continue 7 days off, 7 days on.

While receiving the study treatment, participants will be asked to visit the study site on Day 1 of Cycles 1-8 for tests and procedures. Tests and procedures done for research purposes only include additional blood sample collection and a second fresh research biopsy for biomarker/genetic/immune research.

Participants who benefit from the study treatment may be able to receive additional treatment if they progress after stopping the study treatment.

When participants are taken off the study treatment permanently, they will be asked to return to the study site for an End of Study Treatment visit about 30 days after stopping the study treatment to have tests and procedures done for safety purposes.

Participants who are taken off the study treatment for any reason other than disease progression will continue to have radiological assessments and blood draws every 12 weeks for the first year and every 24 weeks after year 1 until they start a new anti-cancer treatment, disease progression, or the study ends. Participants will continue to be followed for survival and to review any new anti-cancer therapies every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced epithelial ovarian, primary peritoneal or fallopian tube carcinomas.
* Patients must have radiologically documented disease progression from their prior line of therapy.
* Patients must have measurable disease based on RECIST 1.1.
* Have received a front line platinum-based regimen (administered via either IV or IP) following primary or interval debulking surgery with documented disease recurrence.
* Have fulfilled the following additional requirements regarding prior treatments depending on the cohort that the patient is to be enrolled in.
* Eastern Cooperative Group (ECOG) performance status <=1.
* Life expectancy greater than 16 weeks.
* Availability of archival tumor tissue samples. Additional samples may be requested if tumor tissue provided is not adequate for quality and/or quantity as assessed by the laboratory.
* Be willing to provide tumor tissue from a newly obtained core or excisional biopsy prior to start treatment and on day 15 of cycle 1.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* Diagnosis of immunodeficiency or therapy with systemic steroid or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* History of autoimmune disease, such as but not restricted to, rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematous, ankylosing spondylitis, scleroderma, or multiple sclerosis requiring treatment within the last two years. Patients with vitiligo or diabetes are not excluded.
* Patients with history of thyroiditis within 5 years.
* Patients with known history of active TB (Bacillus Tuberculosis).
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Hypersensitivity to Pembrolizumab, DPX-Survivac immunovaccine, Cyclophosphamide or any of their excipients.
* Patients that have received a live vaccine within 30 days of planned start of study therapy.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent or DPX-Survivac vaccine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 5 years
  ORR will be used to evaluate the clinical anti-tumor activity of Pembrolizumab, DPX Survivac and oral cyclophosphamide combination.

SECONDARY OUTCOMES:
Progression free survival (PFS) rate | 5 years
  PFS rate from start of study treatment to time of progression or death whichever comes first
Overall survival (OS) rate | 5 years
  OS rate from start of study treatment until death for every cause
Number of side effects | 5 years
  Adverse events will be analyzed as safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No